CLINICAL TRIAL: NCT02527395
Title: To Determine the Degree of Association Between Heat Pain Detection Threshold and Area of Secondary Hyperalgesia Following Brief Thermal Sensitization in Healthy Male Volunteers
Brief Title: Association Between Heat Pain Detection Threshold and Area of Secondary Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Sejer Hansen, M.D., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: SM2-MSH-2014
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Experimental pain; Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clinical pain models (Other): Brief thermal sensitization. Heat pain detection threshold. Pain during 1 min. thermal stimulation
  Interventions: Other: Brief thermal sensitization; Other: Pain during 1 min. thermal stimulation; Other: Heat pain detection threshold

INTERVENTIONS:
Other: Brief thermal sensitization — A small area of the skin of the study participants are heated to 45 degree celsius for 3 minutes, followed by evaluation of secondary hyperalgesia.
  Other Names: Clinical pain model
Other: Pain during 1 min. thermal stimulation — A small area of the skin of the study participants are heated to 45 degrees celsius for 1 minute. During the 1 minute period, the study participant will continually report pain on an electronic visual analog scale.
  Other Names: Clinical pain model
Other: Heat pain detection threshold — The threshold for heat pain are evaluated by heating a small area of the study participants skin. When the study participant feels pain, the temperature (degrees celsius) is registered. 4 threshold measurements per session. Heat pain threshold is defined as the average temperature of the 4 measurements.
  Other Names: Clinical pain model

SUMMARY:
The purpose of this prospective study is to investigate how close Heat Pain Detection Threshold is associated with the area of secondary hyperalgesia, elicited by the clinical pain model Brief Thermal Sensitization.

Furthermore we wish to investigate how close the clinical pain model: Pain during 1 min. heating of the skin (45 degrees celsius), and the psychological tests, Pain Catastrophizing Scale and Hospital Anxiety and Depression Scale are associated with the area of secondary hyperalgesia, elicited by the clinical pain model Brief Thermal Sensitization.

DETAILED DESCRIPTION:
The study participants will be tested with 3 types of clinical pain models on two separate identical study days. A minimum of 7 days will separate the two study days, thus, the minimum length of the study is 7 days, but can be higher.

The 3 types of pain conditioning consist of 1) Brief thermal sensitisation (BTS), 2) Heat pain detection threshold (HPDT), and pain during 1 min. thermal stimulation (p-TS.

The order of the stimulations (HPDT and BTS) is randomised for each patient and each study day, by a random allocation sequence, computer-generated by Copenhagen Trial Unit and stored in sealed and opaque envelopes to secure adequate allocation concealment. p-TS is conducted subsequent to BTS and HPDT.

The participants will complete the psychological tests Pain Catastrophizing Scale (PCS) and Hospital Anxiety and Depression Scale (HADS) in their private home prior to study day 1. The completed tests will be placed in opaque sealed envelopes to secure blinding of the investigator and outcome assessor.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <35 years
* Speak and understand Danish
* Male gender
* Study participants who have understood and signed the informed consent
* No prescription medicine during the last 30 days.

Exclusion Criteria:

* Study participants that cannot cooperate to the test.
* Study participants who have a weekly intake of >21 units of alcohol, or a have consumed >3 units of alcohol within 24 hours before experimental day.
* Study participants with a substance abuse, assessed by the investigator.
* Study participants, who have consumed analgesics less than 3 days before experimental day.
* Study participants, who have consumed antihistamines less than 48 hours before experimental day.
* Study participants, who have consumed antidepressant medication during the last 30 days before experimental day.
* Study participants with chronic pain.
* Study participants with neurological illnesses.
* Study participants with psychiatric diagnoses.
* Study participants with tattoos on the extremities.
* Study participants with eczema, wounds or sunburns on the sites of stimulation.
* Study participants with a Body Mass Index of >30 kg/m2 or <18 kg/m2

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Size of the Area of secondary hyperalgesia following Brief thermal sensitization, evaluated by cm2, and heat pain detection threshold registered by degrees celsius. | 7 days
  How close is the Heat Pain Detection Threshold associated with the size of the area of secondary hyperalgesia induced by Brief thermal sensitization? Area of secondary hyperalgesia will be investigated on two separate study days separated with a minimum of 7 days. The association will be expressed in R2 and prediction intervals for the area of BTS given fixed values of HPDT.

SECONDARY OUTCOMES:
Pain during 1 min. thermal stimulation, evaluated by Area Under the Curve of the visual analog scale, 0-100 mm. | Study day 1 and 2. A minimum of 7 days
  How close is the Visual analog scale (VAS)-AUC (area under the curve) following pain during 1 min. thermal stimulation associated with the size of the area of secondary hyperalgesia induced by Brief thermal sensitization?
Pain during 1 min. thermal stimulation, evaluated by maximum on the visual analog scale, 0-100mm. | Study day 1 and 2. A minimum of 7 days.
  How close is the max. VAS-score following pain during 1 min. thermal stimulation associated with the size of the area of secondary hyperalgesia induced by Brief thermal sensitization?
Score of Pain Catastrophizing Scale | Study day 1 and 2. A minimum of 7 days.
  How close is the scores of Pain Catastrophizing Scale associated with the size of the area of secondary hyperalgesia induced by Brief thermal sensitization?
Score of Hospital Anxiety and Depression Scale | Study day 1 and 2. A minimum of 7 days.
  How close is the scores of Hospital Anxiety and Depression Scale associated with the size of the area of secondary hyperalgesia induced by Brief thermal sensitization?
Score of Subscales of Pain Catastrophizing Scale and Hospital Anxiety and Depression Scale. | Study day 1 and 2. A minimum of 7 days.
  How close are the subscales in the two psychological tests (PCS-rumination, PCS-magnification, PCS-helplessness, and HADS-Anxiety, HADS-Depression) associated with the size of the area of secondary hyperalgesia?

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anaesthesia and surgery, 4231, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen MS, Asghar MS, Wetterslev J, Pipper CB, Johan Martensson J, Becerra L, Christensen A, Nybing JD, Havsteen I, Boesen M, Dahl JB. Is the Volume of the Caudate Nuclei Associated With Area of Secondary Hyperalgesia? - Protocol for a 3-Tesla MRI Study of Healthy Volunteers. JMIR Res Protoc. 2016 Jun 17;5(2):e117. doi: 10.2196/resprot.5680. PMID 27317630
- [Derived] Hansen MS, Wetterslev J, Pipper CB, Asghar MS, Dahl JB. Is heat pain detection threshold associated with the area of secondary hyperalgesia following brief thermal sensitization? A study of healthy volunteers - design and detailed plan of analysis. BMC Anesthesiol. 2016 May 31;16(1):28. doi: 10.1186/s12871-016-0193-2. PMID 27246322